CLINICAL TRIAL: NCT05111743
Title: Real-world Evaluation of Brolucizumab for the Treatment of Neovascular (Wet) Age-related Macular Degeneration (AMD) (Komodo Health)
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CRTH258AUS21
Record Dates: First submitted 2021-10-22; First posted 2021-11-08 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-12

CONDITIONS: Age-related Macular Degeneration (AMD)
Keywords: Brolucizumab,; intravitreal injection,; neovascular age-related macular degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — brolucizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Brolucizumab: Participants received brolucizumab injection during the index period
  Interventions: Drug: Brolucizumab

INTERVENTIONS:
Drug: Brolucizumab — Participants received brolucizumab injection during the index period
  Other Names: BEOVU®

SUMMARY:
This study was a retrospective cohort study of patients to assess the early insights into real-world safety among wet AMD patients initiating brolucizumab. Evidence was generated to describe their patient characteristics and clinical outcomes. The study was conducted using the Komodo Healthcare Map.

DETAILED DESCRIPTION:
Komodo Healthcare Map claims data from 08-Oct-2016 to the date of most recent data from patients with wet AMD who initiated brolucizumab were analyzed in this study.

* Identification period of the index date (index period): The patients fulfilling the selection criteria were identified during the period from 08-Oct-2019 to 30-Apr-2020.
* Index date: Defined as the date of the earliest brolucizumab injection during the index period.
* Study Period: The period from 08-Oct-2016 to the most recent data extraction date (05-Jun-2020).

  o Note since 05-Jun-2020 was the date data was pulled, claims data from recent months (e.g. May) may be incomplete (relative to the final DB state) as well.
* Pre-index period: The period 36 months prior to the index date

  o Note: Data within 36 months prior to the index date will be used to assess baseline characteristics.
* Post-index period: The period of 180 days after the index date

ELIGIBILITY:
Inclusion criteria:

1. ≥1 Healthcare Common Procedure Coding System (HCPCS) code (J code) or National Drug Code (NDC) for treatment with brolucizumab during the index period (date of earliest code = index date)
2. ≥18 years old on the index date
3. ≥1 International Classification of Diseases, Clinical Modification-9/10 (ICD-9/10) code for wet AMD in the 36 months prior to or on the index date

   * Note: Off-label use of brolucizumab is not expected given payer access restrictions in the US
4. ≥24 months of continuous enrollment prior to the index date
5. ≥1 follow-up visit related to their wet AMD after the index date

Exclusion criteria:

1. Use of brolucizumab prior to 08-Oct-2019 (e.g. clinical trials)
2. Unknown laterality of the index eye on the index date
3. Patients with no data throughout the 12 months immediately prior to the index date

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with wet AMD who initiated brolucizumab were analyzed in this study.
Sampling Method: Non-Probability Sample
Enrollment: 9261 (Actual)
Dates: Start 2020-06-17 (Actual); Primary Completion 2020-12-18 (Actual); Study Completion 2020-12-18 (Actual)

PRIMARY OUTCOMES:
Number of patient eyes with an Intraocular Inflammation (IOI) event during the first 6 months | Up to 6 months post brolucizumab injection
  To assess IOI events observed after starting treatment with brolucizumab

SECONDARY OUTCOMES:
Age | Index date defined as the date of the earliest brolucizumab injection during the index period (from 08-Oct-2019 to 30-Apr-2020)
  Age information was reported
Gender information | Index date defined as the date of the earliest brolucizumab injection during the index period (from 08-Oct-2019 to 30-Apr-2020)
  Gender information was reported
Number of patients at various Patient Region | Index date defined as the date of the earliest brolucizumab injection during the index period (from 08-Oct-2019 to 30-Apr-2020)
  Patient regions: Northeast, Midwest, South, West, Unknown
Number of patients with Insurance type | Index date defined as the date of the earliest brolucizumab injection during the index period (from 08-Oct-2019 to 30-Apr-2020)
  Insurance type: Private, Medicare, Medicare Advantage, Medicaid, Other
Number of patients with Laterality of wet Age-related macular degeneration (AMD) | Index date defined as the date of the earliest brolucizumab injection during the index period (from 08-Oct-2019 to 30-Apr-2020)
  Laterality of wet AMD: Unilateral, Bilateral
Number of patients with Laterality of any Age-related macular degeneration (AMD) | Index date defined as the date of the earliest brolucizumab injection during the index period (from 08-Oct-2019 to 30-Apr-2020)
  Laterality of wet AMD: Unilateral, Bilateral
Number of eyes with the concurrent eye disease | Within 180 days prior to the index date (inclusive of the index date) ( index date defined as the date of first brolucizumab injection)
  Types of concurrent eye diseases:
  * Cataracts
  * Posterior vitreous detachment
  * Puckering of macula
  * Macular hole
  * Vitreomacular traction
  * Glaucoma
  * Amblyopia
  * Papillitis
  * Ischemic optic atrophy
  * Diabetic retinopathy
  * Diabetic macular edema
  * Hypertensive retinopathy
  * Pathologic myopia
  * RAO
  * RO
  * RV
  * Vitritis
  * Endophthalmitis
  * Uveitis
  * Choroidal neovascularization (due to causes other than AMD, if possible, to determine)
  * IOI
Number of patient eyes with previous ocular surgeries or procedures | Within 180 days prior to the index date (inclusive of the index date) ( index date defined as the date of first brolucizumab injection)
  Types:
  * Laser photocoagulation (or laser therapy)
  * Photodynamic therapy (PDT)
  * Glaucoma surgery (trabeculectomy, MIGS)
  * Cataract surgery
  * Iridotomy
  * Ocular radiation
  * Panretinal photocoagulation
  * Submacular surgery, other surgical intervention or laser treatment for AMD
  * Vitrectomy
  * Scleral buckle
  * Pneumatic retinopexy
  * Cryopexy
Number of patient eyes with systemic comorbidities | 36-month period prior to the index date (inclusive of the index date) ( index date defined as the date of first brolucizumab injection)
  Types:
  * Obesity
  * Cerebrovascular disease
  * Peripheral vascular disease
  * Diabetes
  * Renal disease
  * Chronic pulmonary disease
  * Congestive heart failure
  * Any malignancy, including lymphoma and leukemia
  * Myocardial infarction
  * Dementia
  * Arteriothrombotic event
  * Thromboembolytic event
  * Atherosclerosis
  * Arterial hypertension
  * Ischemic heart disease
  * Atrial fibrillation
  * Lipid disorders
  * Cardiac septal defect
  * Valvular cardiac defect
  * Hyperlipidemia
  * Hypercholesterolemia
  * Atherosclerotic disease
  * Thrombosis
  * Carotid artery disease
Number of Concomitant systemic medications (chronic use) | 36-month period prior to the index date (inclusive of the index date) ( index date defined as the date of first brolucizumab injection)
  Types:
  * Corticosteroids
  * Systemic anti-VEGFs
  * Lipid lowering agents
  * Antihypertensives
  * Biologics
  * Antimetabolites/cancer therapy
  * Anticoagulants
Number of patient eyes with the Cataract status | 36-month period prior to the index date (inclusive of the index date) ( index date defined as the date of first brolucizumab injection)
  Types: phakic, pseudophakic, aphakic
Number of patient eyes with Intraocular inflammation | 12 and 6 months prior to the index date (inclusive of the index date) ( index date defined as the date of first brolucizumab injection)
  The following categories were reported:
  * No history of IOI and endophthalmitis related to safety evaluation and panuveitis
  * History of IOI and endophthalmitis related to safety evaluation and panuveitis
  * History of IOI including panuveitis (excluding endophthalmitis related to safety evaluation)
  * History of endophthalmitis related to safety evaluation
  * History of panuveitis
Number of patient eyes with the history of ocular inflammation (includes IOIs or panuveitis or endophthalmitis relevant to safety evaluation) | 36-month period prior to the index date (inclusive of the index date) ( index date defined as the date of first brolucizumab injection)
  The following categories were reported:
  * History of anterior inflammation
  * History of posterior inflammation
  * No history of IOI or endophthalmitis related to safety evaluation or panuveitis
  * History of IOI and/or endophthalmitis related to safety evaluation and/or panuveitis
  * History of IOI including panuveitis (excluding endophthalmitis related to safety evaluation)
  * History of endophthalmitis related to safety evaluation
  * History of Panuveitis
History of other IOI and endophthalmitis due to infections or other underlying disease | 36, 12 and 6 months prior to the index date (inclusive of the index date) ( index date defined as the date of first brolucizumab injection)
  The following categories were reported:
  * No history of inflammation
  * History of any ocular inflammation
  * History of severe ocular inflammation
  * History of anterior inflammation
  * History of posterior inflammation
  * History of IOI or endophthalmitis due to infections and other underlying disease (separate category)
Number of patient eyes with prior Intraocular Inflammation (IOI) and/or prior Retinal vascular occlusion (RO) | 12 months prior to the index date ( index date defined as the date of first brolucizumab injection)
  Included history of ocular inflammation or occlusion
Number of patient eyes with Systemic inflammation / auto-immune history (in total and at the event level) | 36-month period prior to the index date (inclusive of the index date) ( index date defined as the date of first brolucizumab injection)
  The following categories were reported:
  * Systemic vasculitis
  * Rheumatoid arthritis
  * SLE
  * Multiple sclerosis
  * Sarcoidosis
  * Giant cell arteritis / Temporal arteritis
  * HLA-B27 diseases
  * Behcet/Behcet's disease
  * Ankylosing Spondylitis
  * Crohn Disease
  * Drug Hypersensitivity
  * Vogt-Koyanagi-Harada (VKH)
Number of patient eyes with the Provider specialty | Index date defined as the date of the earliest brolucizumab injection during the index period (from 08-Oct-2019 to 30-Apr-2020)
  The following types were included:
  Retina specialist, General ophthalmologist, Non-retina specialist, unknown
Number of patient eyes with Concomitant ocular medications | 36-month period prior to the index date (inclusive of the index date) ( index date defined as the date of first brolucizumab injection)
  The following types were included: any corticosteroids [prednisone, prednisolone acetate, difluprednate, Kenalog, ozurdex, yutiq], biologics [adalimumab], cyclosporine, azathioprine, methotrexate, ganciclovir, acyclovir, valacyclovir, foscavir, trifluridine, mycophenolate, rituxan, vancomycin, prostaglandins
Type of exam performed | 30 days before or on first brolucizumab injection (index date)
  OCT, FA, CP - color photo or color fundus photo
Number of eyes treated with brolucizumab | Index date defined as the date of the earliest brolucizumab injection during the index period (from 08-Oct-2019 to 30-Apr-2020)
  The following types were included:
  OD [eye, right], OS [eye, left], Unspecified, Unilateral, Bilateral)
Number of patient eyes with Anti-VEGF treatment-naive vs prior-treated | 60 months prior to index ( index date defined as the date of first brolucizumab injection)
  Anti-VEGF treatment-naive vs prior-treated were measured at the eye-level
Number of patient eyes with prior treatment status | 60 months prior to index ( index date defined as the date of first brolucizumab injection)
  The following types were included: off-label bevacizumab, ranibizumab, aflibercept, unknown, treatment-naive
Number of patient eyes with different prior anti-VEGF agents | 60 months prior to index ( index date defined as the date of first brolucizumab injection)
  Following categories will be included : 0, 1, 2, ≥3
Number of patient eyes with prior anti-VEGF agents (total, per anti-VEGF agent) | 60 months prior to index ( index date defined as the date of first brolucizumab injection)
  Following categories will be included :
  * Continuous
  * Categorical: <6, 6 to <12, 12 to <24, ≥24
Number of patient eyes with the Last injection inetrval | 60 months prior to index ( index date defined as the date of first brolucizumab injection)
  Following categories will be included :
  * Continuous (weeks)
  * Categorical: <4, 4 to <6, 6 to <8, ≥8, <12, ≥12 weeks
Duration of last anti-VEGF treatment (total, per anti-VEGF agent) | 60 months prior to index ( index date defined as the date of first brolucizumab injection)
  Following categories will be included :
  * All anti-VEGFs i. Continuous ii. Categorical: <6, 6 to <12, 12 to <24, ≥24 months
  * Specific anti-VEGF iii. Continuous (days)
Time since wet Age-related macular degeneration (AMD) diagnosis | 36-month period prior to the index date (inclusive of the index date) ( index date defined as the date of first brolucizumab injection)
  Patients were measured at the eye level
Time since any Age-related macular degeneration (AMD) diagnosis | 36-month period prior to the index date (inclusive of the index date) ( index date defined as the date of first brolucizumab injection)
  Patients were measured at the eye level
Time from last anti-VEGF injection to index date | 60 months prior to index ( index date defined as the date of first brolucizumab injection)
  The following categories were measured:
  * Continuous (days)
  * Categorical (0-30, 31-60, 61-90, 91+ days)
Number of ocular adverse events (AEs) | Post-index period defined as the 180 days following therapy initiation, excluding index date
  To assess the incidence of ocular AEs among patients treated with brolucizumab

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, East Hanover, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Results for CRTH258AUS21 from the Novartis Clinical Trials Website — http://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17875